CLINICAL TRIAL: NCT00606333
Title: A Randomized, Multi-Center, Single-Blind Comparison of the Conor Cobalt Chromium Reservoir Based Stent With Sirolimus Elution Versus the TAXUS Liberte Paclitaxel-eluting Coronary Stent System in De Novo Native Coronary Artery Lesions
Brief Title: Comparison of the Conor Sirolimus-eluting Coronary Stent to the Taxus Liberte Paclitaxel-eluting Coronary Stent in the Treatment of Coronary Artery Lesions
Acronym: NEVO RES-I
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The NEVO™ stent will not be commercialized. Cordis have decided to close the study after 3 years. This decision took the absence of safety signals into account.
Sponsor: Cordis US Corp. (Industry)
Collaborators: Conor Medsystems (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP-06
Record Dates: First submitted 2008-01-17; First posted 2008-02-01 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Coronary Atherosclerosis
Keywords: Coronary artery disease; drug-eluting stents; sirolimus-eluting coronary stents
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Investigational arm (Experimental): Subjects randomized to treatment with the NEVO™ Sirolimus-eluting Coronary Stent System.
  Interventions: Device: NEVO™ Sirolimus-eluting Coronary Stent System
- Control Arm (Active Comparator): Subjects randomized to treatment with the TAXUS Liberte Paclitaxel-eluting Coronary Stent System.
  Interventions: Device: Drug-eluting stent (TAXUS Liberte Paclitaxel-eluting Coronary Stent System)

INTERVENTIONS:
Device: NEVO™ Sirolimus-eluting Coronary Stent System — Intervention will consist of percutaneous coronary intervention for treatment of a single coronary lesion using standard coronary intervention techniques. Intervention in this arm will include treatment with the Conor Cobalt Chromium Sirolimus-eluting Coronary Stent System. Subjects assigned to the IVUS sub-study population will undergo intravascular ultrasound evaluation immediately post-stenting.
  Arms: Investigational arm
Device: Drug-eluting stent (TAXUS Liberte Paclitaxel-eluting Coronary Stent System) — Intervention will consist of percutaneous coronary intervention for treatment of a single coronary lesion using standard coronary intervention techniques. Intervention in this arm will include treatment with the TAXUS Liberte Paclitaxel-eluting Coronary Stent System. Subjects assigned to the IVUS sub-study population will undergo intravascular ultrasound evaluation immediately post-stenting.
  Other Names: Taxus Liberte Paclitaxel-eluting Coronary Stent System
  Arms: Control Arm

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the Conor Sirolimus-eluting Coronary Stent System in the treatment of coronary artery disease (a single atherosclerotic lesion) in native coronary arteries. The study will evaluate the outcomes of a new drug-eluting stent compared to an approved drug-eluting stent.

While Cordis made a business decision to no longer pursue NEVO™ development and commercialization, the patients will be followed up as per protocol. This includes performing all protocol required follow-up visits and the collection and reporting of all safety information.

DETAILED DESCRIPTION:
Restenosis remains a frequent cause of late failure following successful coronary angioplasty occurring in an estimated 20-40% of procedures performed. Coronary stents provide mechanical scaffolding that helps reduce restenosis by limiting the extent of elastic recoil and late vascular remodeling. Despite improvements over balloon angioplasty alone, restenosis following coronary stenting procedures has been cited to occur in 20-40% of cases and is primarily a result of neointimal hyperplasia. Thus, stents which are capable of delivering drugs to limit neointimal hyperplasia, in addition to providing mechanical support at the area of the lesion, have been developed to further limit the extent of restenosis following coronary stenting. There are several pharmacologic agents approved for use with drug-eluting stents.Two drugs have been widely studied in controlled clinical trials and real-world patient populations, sirolimus and paclitaxel.

This study will evaluate a new sirolimus-eluting cobalt chromium coronary stent system compared to an approved paclitaxel-eluting coronary stent system in the treatment of single de novo coronary lesions in native coronary arteries. Subjects meeting qualification will be randomized in a 1:1 fashion to treatment with the Conor sirolimus-eluting coronary stent or to treatment with an approved paclitaxel-eluting coronary stent. All subjects will undergo angiographic follow-up at six months and complete clinical follow-up for a period of five years.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Eligible for percutaneous coronary intervention and coronary artery bypass graft surgery.
* Diagnosis of stable or unstable angina or silent ischemia
* Left ventricular ejection fraction >30%
* The subject requires treatment of a single de novo lesion in a native coronary artery.
* Lesion to be treated is less than or equal to 28 mm in length in a vessel that is 2.5-3.5mm diameter.
* The target lesion diameter stenosis is >50% and <100% by visual estimate.
* The target lesion is a minimum of 10 mm distance from any previously treated segment of the target vessel.
* The subject understands the study requirements, is willing to comply with all study procedures and has provided written informed consent.

Exclusion Criteria:

* The subject has undergone coronary revascularization to any vessel within 30 days.
* The subject has undergone target vessel revascularization within 6 months.
* Treatment of more than one qualifying lesion is required at the time of enrollment, or is planned within 30 days following enrollment.
* The subject has known sensitivity to sirolimus, paclitaxel, the polymeric matrices, stainless steel or cobalt chromium.
* There is planned treatment of the target lesion with any device other than the pre-dilatation balloon angioplasty catheter.
* The subject had a myocardial infarction within 72 hours, or presents with CK elevation > 2 times upper limit normal associated with elevated CK-MB.
* The subject is in cardiogenic shock.
* The subject had a cerebrovascular accident within the past 6 months.
* The subject has acute or chronic renal dysfunction (defined as creatinine >2.0 mg/dl).
* The subject has a contraindication to aspirin or clopidogrel.
* The subject has thrombocytopenia (platelet count < 100,000/mm3.
* The subject has had active gastrointestinal bleeding within the past 3 months.
* The subject has a known bleeding or hypercoagulable disorder.
* The subject has had prior anaphylactoid reaction to contrast agents or has contrast sensitivity that cannot be controlled with pre-medication.
* The subject is currently taking immunosuppressant therapy.
* The subject is currently, or has been treated wtih either Rapamune or paclitaxel within 12 months of the procedure.
* The subject is a female with a positive pregnancy test or is lactating.
* The subject has an active infection.
* The subject has co-morbidities that could interfere wtih completion of study procedures, or life expectancy less than 24 months.
* The subject is participating in another investigational drug or device trial that has not completed the primary endpoint or would interfere with the endpoints of this study.

Angiographic Exclusion Criteria

* Left main disease >50% diameter stenosis.
* The target lesion is ostial.
* The target lesion or target vessel are severely calcified.
* The target lesion involves a bifurcation with diseased branch vessel greater than or equal to 2.0 mm that would require intervention or protection.
* The target lesion has TIMI o or TIMI I flow.
* Angiographic evidence of thrombus.
* The target vessel has had prior stent placement.
* The patient has had prior coronary brachytherapy.
* There is angiographic restenosis of any previously treated segment of the target vessel, or atherosclerotic area wtih >50% diameter stenosis outside of the target lesion.
* The subject has undergone prior CABG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2008-03; Primary Completion 2009-05 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Angiographic endpoint of in-stent late lumen loss as measured by QCA. | 6 months

SECONDARY OUTCOMES:
Target Lesion Failure defined as cardiac death that cannot be clearly attributed to a non-cardiac event or non-target vessel, target vessel related myocardial infarction or clinically driven target lesion revascularization. | hospital discharge, 30 days, 6 months and annually through five years.
Target Vessel Failure defined as any myocardial infarction or cardiac death that cannot be attributed to a non-target vessel or any target vessel revascularization. | Hospital discharge, 30 days, 6 months and annually through five years
Major Adverse Cardiac Events defined as an adjudicated composite of death, emergent coronary artery bypass graft surgery, target lesion revascularization, or new myocardial infarction. | Hospital discharge, 30 days, 6 months and annually through five years
Incidence of stent thrombosis | Hospital discharge, 30 days, 6 months and annually through five years
Incidence of target lesion revascularization and target vessel revascularization. | Hospital discharge, 30 days, 6 months and annually through five years
Device Success | Procedural
Lesion success | Procedural
Procedure Success | Hospital Discharge
Angiographic in-stent and in-segment binary restenosis. | 6 months
In-stent minimum lumen diameter | 6 months
Percent volume obstruction of the stent by intravascular ultrasound evaluation | 6 months
Patient reported outcomes as measured by three standardized quality of life surveys. | Baseline, 30 days, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: John Ormiston, MB ChM, Principal Investigator — Mercy Angiography Unit; Alexandre Abizaid, MD. PhD, Principal Investigator — Instituto Dante Pazzanese de Cardiologia
Locations (2):
- Instituto Dante Pazzanese de Cardiologia, São Paulo, Brazil
- Mercy Angiography Unit, Epsom, Auckland, New Zealand

REFERENCES:
- [Result] Ormiston JA, Abizaid A, Spertus J, Fajadet J, Mauri L, Schofer J, Verheye S, Dens J, Thuesen L, Dubois C, Hoffmann R, Wijns W, Fitzgerald PJ, Popma JJ, Macours N, Cebrian A, Stoll HP, Rogers C, Spaulding C; NEVO ResElution-I Investigators. Six-month results of the NEVO Res-Elution I (NEVO RES-I) trial: a randomized, multicenter comparison of the NEVO sirolimus-eluting coronary stent with the TAXUS Liberte paclitaxel-eluting stent in de novo native coronary artery lesions. Circ Cardiovasc Interv. 2010 Dec;3(6):556-64. doi: 10.1161/CIRCINTERVENTIONS.110.946426. Epub 2010 Nov 9. PMID 21062998
- [Result] Otake H, Honda Y, Courtney BK, Shimohama T, Ako J, Waseda K, Macours N, Rogers C, Popma JJ, Abizaid A, Ormiston JA, Spaulding C, Cohen SA, Fitzgerald PJ. Intravascular ultrasound results from the NEVO ResElution-I trial: a randomized, blinded comparison of sirolimus-eluting NEVO stents with paclitaxel-eluting TAXUS Liberte stents in de novo native coronary artery lesions. Circ Cardiovasc Interv. 2011 Apr 1;4(2):146-54. doi: 10.1161/CIRCINTERVENTIONS.110.957175. Epub 2011 Mar 8. PMID 21386089
- [Derived] Abizaid A, Ormiston JA, Fajadet J, Mauri L, Schofer J, Verheye S, Dens J, Thuesen L, Macours N, Qureshi AC, Spaulding C; NEVO ResElution-I Investigators. Two-year follow-up of the NEVO ResElution-I(NEVO RES-I) trial: a randomised, multicentre comparison of the NEVO sirolimus-eluting coronary stent with the TAXUS Liberte paclitaxel-eluting stent in de novo native coronary artery lesions. EuroIntervention. 2013 Oct;9(6):721-9. doi: 10.4244/EIJV9I6A116. PMID 23518218